CLINICAL TRIAL: NCT04348864
Title: Assessment of COVID-19 Diagnostic Self-testing Using Virtual Point-of-care
Brief Title: COVID-19 Diagnostic Self-testing Using Virtual Point-of-care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuroganics LLC (Industry)
Collaborators: Neuroganics Diagnostics LLC (Unknown); Artron Laboratories Inc (Unknown); AllBio Science Inc. (Unknown); Turklab (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/03/18
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Communicable Disease; COVID-19; Sars-CoV2; Infectious Disease; Coronavirus; Virus
Keywords: COVIDscanDX; Antigen test; LAMP test; Diagnostic reader
MeSH Terms: conditions — Communicable Diseases; COVID-19; Coronavirus Infections; Virus Diseases | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Subject with or without symptoms consistent with COVID-19 and have been tested at the point of care (POC) with a molecular diagnostic test (e.g. PCR or isothermal LAMP) or clinical diagnosis, and have been determined to be positive or negative will undergo testing for antibodies or antigen or viral RNA. Roughly three times more subjects testing negative for SARS-CoV-2 compared to positive subjects are expected to be tested from NP samples gathered at the POC by POC staff or self-swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Positive-Antigen swab test for SARS-COV-2 (Experimental): Subjects who have tested positive for the presence of SARS-COV-2 viral antigen using a rapid test or LAMP/PCR-based molecular test from nasal pharyngeal self-swab or a swab administered in a clinical setting at the point of care by a trained clinician. Parallel PCR-based testing occurs in an advanced laboratory to obtain Ct values for positive test results.
  Interventions: Diagnostic Test: COVID-19 Antigen/Antibody Rapid Testing, mobile device image capture and telemedicine support; Other: Telemedicine
- Negative-Antigen swab test for SARS-COV-2 (Sham Comparator): Subjects who have tested negative for the presence of SARS-COV-2 viral antigen using a rapid test or LAMP/PCR-based molecular nasal pharyngeal self-swab or a swab administered in a clinical setting by a trained clinician. PCR-based testing occurs in an advanced laboratory.
  Interventions: Diagnostic Test: COVID-19 Antigen/Antibody Rapid Testing, mobile device image capture and telemedicine support; Other: Telemedicine

INTERVENTIONS:
Diagnostic Test: COVID-19 Antigen/Antibody Rapid Testing, mobile device image capture and telemedicine support — An immunodiagnostic rapid (5-20 minute) test detects circulating antibodies in the blood, serum or plasma of individuals who have been infected with the novel coronavirus SARS-COV-2 as detected by rapid antigen test or LAMP/PCR-based molecular test taken from nasopharyngeal swab samples in the recent past.
  Other Names: COVID-19 diagnostic rapid testing reader and software validation
Other: Telemedicine — Imaging of the test using the software application COVIDscanDX and upload to server by the subject and phone, video or messaging consult with a clinician for interpretation and instructions establishes the telemedicine (i.e. virtual point-of-care).
  Other Names: virtual point-of-care

SUMMARY:
The goal of the research is to assess candidate COVID-19 rapid diagnostic tests (e.g. immunodiagnostic antibody tests, like Cellex qSARS-CoV-2 IgG/IgM Rapid Test, or antigen tests, like Turklab Test-It COVID-19 Home Test, AllBio Science Inc. and Artron Laboratories Inc. rapid COVID-19 antigen tests in order to judge their clinical accuracy compared to Centers for Disease Control (CDC)-recommended molecular genetic testing and clinical diagnosis. Second, it is our goal to determine if self-testing assisted by COVIDscanDX mobile device camera acquisition software platform and telemedicine clinical/technical support (virtual point-of-care) improves the ease of use and immediate interpretation of the tests, thus making self-testing comparable in accuracy and safety to testing in a clinical setting. Third, we are testing antibodies to SARS-CoV-2 after diagnosis with COVID-19 or following vaccination to measure the onset and time course of detectable antibodies from finger-stick blood drops and rapid antibody lateral flow tests. The overall purpose of the study is to dramatically increase the capacity of COVID-19 testing by establishing the safety, ease-of-use and validity of self-testing assisted by mobile device imaging and telemedicine remote support and provide evidence of antibody time-course response to vaccination.

DETAILED DESCRIPTION:
Two Nasopharyngeal (NP) swabs will be collected from opposite nares by health care professionals at the POC from minimally 500 subjects enrolled at a minimum of 2 point- of-care (POC) clinical sites. One swab will be tested for the presence of SARS-CoV-2 responsible for COVID -19 using antigen-based tests. A second swab will be placed in transport media and transferred to a laboratory for testing using a high sensitivity EUA real-time (RT) PCR assay as the comparator method and the Ct values used to determine positive or negative. The order of sample collection will be randomized.

Serial testing for home use of the Test-It (Turklab) COVID-19 Rapid Antigen test will be tested in symptomatic and asymptomatic subjects.

Positive tests will be tested for SARS-CoV-2 variant using Whole Genome Sequencing Method by Amplicon-Based NGS (Quest Diagnostics).

Two to 4 health care professional operators per site, with a range of education and training, at a point of care setting will perform a COVID-19 Rapid test assay utilizing the Instructions for Use and/or Quick Reference Instruction.

Sample Population: Males and females, age 2 and older, with or without symptoms consistent with SARS-CoV-2 infection (COVID-19).

Outcome measures: 1) Sensitivity and specificity will be calculated for comparison of results between the Rapid test and the high sensitivity EUA real-time (RT) PCR assay comparator. 2) Evidence that a Health Care Professional (HCP) at Point of Care (POC) can safely and effectively utilize the Rapid test and the COVIDscanDX reader after reading the Instructions For Use (IFU) and/or brief instruction video.

Antibody testing will be performed after PCR/antigen testing or after vaccination with and FDA EUA allowed SARS-CoV-2 vaccine. A finger-stick blood drop, nasopharyngeal swab or saliva sample in buffer is applied to a lateral flow test to measure either SARS-CoV-2 antigen or IgM and IgG antibodies either once or up to five times separated by a week for 35 days after vaccination. Follow-up tests may be performed to measure the longevity of the antibody response over time up to a year.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have experienced symptoms of COVID-19 and have been tested using a CDC approved or FDA registered and listed nucleic acid based test within 1 year of Feb 1, 2020.
* Individuals who have been clinically diagnosed or suspected to have had COVID-19.
* Individuals who are at the time of enrollment in the study currently or in the recent past (3 weeks) exhibiting symptoms of COVID-19.
* Individuals capable of performing a finger stick blood drop draw or saliva collection and placing it in a sample collection tube.
* Individuals that have interacted with a COVID-19 positive individual and are still exhibiting symptoms will be tested by a CDC approved or FDA registered nucleic acid based device.
* Individuals must be capable of navigating a mobile device to take an image of the test using the camera and enter information into fields on the device and wireless/cellular capability to upload one or more images to a website server.

Exclusion Criteria: Individuals incapable of pricking their finger and placing a drop of blood into a sample well.

* Individuals who cannot navigate a mobile device and see the screen to navigate and enter information in fields or align the camera with the test image.
* Pregnant woman are not excluded if they meet the inclusion criteria and age requirements.
* Individuals with a deviated septum
* Cognitively impaired individuals resulting in the inability to provide informed consent,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Clinical accuracy of the antibody and antigen rapid tests compared to LAMP/PCR-based test result | 1 year
  Accuracy refers to the amount of agreement between the results of the antibody-based rapid test and the results of a PCR-based reference test
Clinical accuracy of the antibody and antigen rapid tests based on Clinical diagnosis | 1 year
  Accuracy refers to the amount of agreement between the results of the rapid tests and a clinical diagnosis of COVID-19
Self-test interpretation of result vs expert clinical image interpretation of result | 1 year
  Clinical accuracy of the subject's visual interpretation of the test result vs image analysis from clinician

SECONDARY OUTCOMES:
Ease of self-testing procedure | 1 year
  Subjects will complete a survey to rate the testing procedure for ease of use and convenience. The survey will ask subjects to rate the ease of use on a scale from 1 (easiest procedure to complete and understand) to 10 (most complicated and confusing procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Cooper, Ph.D., Principal Investigator — Neuroganics LLC
Locations (1):
- Neuroganics, Northglenn, Colorado, United States

IPD SHARING:
Plan to Share IPD: No